CLINICAL TRIAL: NCT05786898
Title: NEAR-TSA : Adaptation of the NEAR (Neuropsychological and Educational Approach of Cognitive Remediation) Cognitive Remediation Method to Child and Adult Autism by Including Social Scenarios and Skills
Brief Title: Adaptation of the NEAR Cognitive Remediation Method to Child and Adult Autism by Including Social Scenarios and Skills
Acronym: NEAR-TSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D22-P018
Record Dates: First submitted 2022-12-13; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Cognitive remediation; Children; Adults
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEAR TSA (Experimental): Neuropsychological and Educational Approach of Cognitive Remediation, adapted for autism (NEAR-TSA)
  Interventions: Other: NEAR-TSA

INTERVENTIONS:
Other: NEAR-TSA — Neuropsychological and Educational Approach of Cognitive Remediation adapted to autism
  32 sessions spread over 4 to 8 months (1 session per week for minors, 2 sessions per week for adults), lasting 90 to 120 minutes

SUMMARY:
The investigators currently provide the NEAR method (neuropsychological educational approach to cognitive remediation) for people with neurocognitive difficulties, without distinguishing between ASD and schizophrenia.

However, the NEAR method does not address social cognition in the stimulated functions. The aim of this study is to add social scenarios to this neurocognitive method in order to improve not only neurocognitive functions, but also social cognition. Thus, NEAR would be in this adapted form a method that could be completely adapted to autism spectrum disorders in preadolescents and adults.

The study will include participants aged 13-40 years, with a diagnosis of ASD.

The NEAR TSA method will include 32 sessions:

* one session (90-120 min, with one or two breaks) per week for 32 weeks (8 months), for minor participants.
* two sessions (90 minutes each, with no breaks) per week for 16 weeks (4 months), for adult participants.

The method includes 30 minutes of computerized exercises, 15 minutes of discussion on the exercises performed and the strategies applied, and the rest of the time for "bridging groups".

Three evaluation are proposed:

* an initial clinical and functional evaluation (T1), before the beginning of the program,
* a second clinical, functional and neuropsychological evaluation (T2), within one month since the end of the program
* a third clinical, functional and neuropsychologica evaluationl (T3), three months after the end of the program.

DETAILED DESCRIPTION:
Inclusion age:two samples: 13 to 15 years old and 16 to 40 years old the clinical evaluation (T1,T2, T3) includes: global functional assessment; questionnaires for children and adults including the self esteem questionnaire, quality of life (who_QOL Bref), social responsiveness scale, conversational skills (CCC-2 for children; Pomini Scale for adults), intrinsic motivational scale (Medalia), Satisfaction scale (CSQ8).

The Neuropsychological evaluation (T1, T2, T3) includes: WISC5 (children), WAIS 4 (adults), stroop test, D2-R, Child memory scale or Wechsler Memory scale for adults, Brief, color trail test, verbal fluency.

Near TSA is a group cognitive remediation method, including one weekly session for children or 2 weekly sessions for adults with 30 mn of neuropsychological exercices, 15 mn of discussion about exercices and strategies, and 30 mn of bridging groups including social scritps.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis Autism Spectrum Disorder (ASD) - (DSM5)
* Attending one of the outpatient units participating in the research
* Diagnosis confirmed by the ADI (Autism Diagnostic Interview) with at least one parent present; or by the ADOS (Autism Diagnosis Observation Schedule)
* Score of at least 7 on the WISC5 (children) or WAIS4 (adults) comprehension subtest
* Patient whose neuropsychological evaluation shows neurocognitive impairment as assessed by the neuropsychologist
* Level of comprehension and communication allowing to understand the instructions of the exercises presented on the screen.
* For children, persons who can attend a non-specialized school
* If the patient is being treated with a psychotropic drug: stability of treatment for more than one month.

Exclusion Criteria:

* Previously known diagnosis of intellectual disability
* Misunderstanding of questions or instructions given during the diagnostic interview
* Proven neurological pathology
* Persons treated with electroconvulsive therapy within the last 6 months
* Uncorrected sensory perception disorder
* Patient participating in another research study with an exclusion period still in progress at inclusion
* Treatment with daytime anxiolytics, and treatment with anticholinergic correctors
* Pregnant or breastfeeding woman
* Participants who have had cognitive remediation in the last two years

Specific exclusion criteria for the "adult" group:

- heterogeneous levels of development highlighted in the diagnostic workup including an examination of cognitive functions

Specific exclusion criteria for the "children" group:

- out-of-school children

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Compliance | At the end of the intervention (Month 4 for adults participants, Month 8 for minor participants)
  number of sessions correctly completed/number of sessions planned
Enrollment rate | at the end of the inclusion period (up to 24 months after the start of the research)
  number of subjects recruited/number of subjects selected
Retention rate | At T2 (between Mont 4 and Month 5 for adults participants ; between Month 8 and Month 9 for minor participants)
  Number of subjects in post evaluation (T2)) / number of subjects recruited

SECONDARY OUTCOMES:
Neuropsychological assessment: attentional performance | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  D2-R test
Neuropsychological assessment : processing speed | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  D2 test
Neuropsychological assessment : flexibility (1) | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the session
  Color Trail Test (raw score)
Neuropsychological assessment : flexibility (2) | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the session
  verbal fluency test (raw score and z-score)
Neuropsychological assessment : flexibility (3) | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the session
  Stroop test (raw score and z-score)
Neuropsychological assessment : working memory | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  Child memory scale for minor <16 years, Wechsler's memory scale for other participants
Functional assessment: quality of life | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  World Health Organization Quality of Life-BREF (WHO QOL-BREF) (26 items rated on a 5-level scale (score from 1 to 5))
Functional assessment : conversational skills | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  CCC-2 (Children's Communication Check list) for minors <16 years (Raw Score, Scaled Score, Percentile)
Functional assessment : conversational skills (2) | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  Pomini's Conversational Skills Scale (1999) for other participants (16 items, score from 0 to 3 for each ; maximum total score : 48)
Functional assessment: self-esteem | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  Rosenberg's Self-Esteem Scale (10 items, score from 1 to 4 for each - total score between 10 and 40)
Functional assessment: global functioning | before the start of the NEAR TSA sessions, within one month of the end of the sessions and 3 to 4 months after the end of the sessions
  Global assessment of functioning scale (total score between 0 and 100)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Amado, Principal Investigator — GHU Paris Saint-Anne
Locations (1):
- GHU Paris Saint-Anne, Paris, France